CLINICAL TRIAL: NCT04829058
Title: A Retrospective and Long-Term Prospective Post Market Clinical Follow-up (PMCF) Study of the GYNECARE GYNEMESH® PS Nonabsorbable PROLENE® Soft Mesh
Brief Title: GYNEMESH PS Mesh Post Marketing Clinical Follow-Up Study
Status: Recruiting | Type: Observational
Sponsor: Ethicon, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: ESC_2020_02
Record Dates: First submitted 2021-03-19; First posted 2021-04-02 (Actual); Last update posted 2026-01-16 (Actual); Status verified 2026-01

CONDITIONS: Pelvic Organ Prolapse
Keywords: GYNECARE GYNEMESH® PS Nonabsorbable PROLENE® Soft Mesh; POP
MeSH Terms: conditions — Pelvic Organ Prolapse | interventions — Methods

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

INTERVENTIONS:
Device: Intervention — There is no intervention, beyond necessary clinical care, in this study. The surgical procedures that were performed in subjects within this study are identical to the surgical procedures the subjects would have received as part of SOC.

SUMMARY:
The objective of this retrospective and prospective, single-arm, observational, multicenter, post-market study is to evaluate outcomes in women who underwent surgery for vaginal or uterine prolapse with a GYNEMESH PS Mesh.

ELIGIBILITY:
Inclusion Criteria:

Subjects who satisfy all of the following criteria will be considered eligible for enrollment in this study:

1. Female subjects who had laparotomic or laparoscopic abdominal sacrocolpopexy, including robotic-assisted, for apical vaginal or uterine prolapse
2. GYNEMESH PS Mesh was used as a bridging material according to the IFU.
3. Able and willing to participate in follow-up
4. Subject or authorized representative has signed the approved informed consent

Exclusion Criteria

Subjects meeting any of the following criteria will be considered not eligible for enrollment in this study:

1. Subjects < 21 years of age at the time of informed consent
2. Subjects who had transvaginal approach for surgery
3. Had undergone a uterus-sparing procedure (sacrohystero or sacrocervicopexy)

Min Age: 21 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Female subjects ≥ 21 years of age
Study Population: Female subjects ≥ 21 years of age:
  * with a baseline diagnosis of apical vaginal or uterine prolapse;
  * who had laparotomic or laparoscopic sacrocolpopexy, including robotic-assisted, for apical vaginal or uterine prolapse within 7 years of enrolment;
  * where GYNEMESH PS Mesh was used as a bridging material, and;
  * who are willing and able to participate in prospective follow-up.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2021-11-24 (Actual); Primary Completion 2031-09-30 (Estimated); Study Completion 2032-03-31 (Estimated)

PRIMARY OUTCOMES:
Physical examination with Pelvic Organ Prolapse Quantification (POP-Q) Assessment CHange | Post-surgery through study completion, approximately 7 yrs
  Objective cure of vaginal or uterine prolapse approximately 7 years after surgery, defined as POP-Q stage ≤2 at point C as determined with physical exam.

SECONDARY OUTCOMES:
Patient Global Impression of Improvement (PGI-I) or Patient Global Impression of Change (PGI-C) Questionnaire | Post-surgery through study completion, approximately 7yrs
Pelvic Floor Distress Inventory (PFDI-20) Questionnaire | Post-surgery through study completion, approximately 7yrs
Pelvic Organ Prolapse/Urinary Incontinence Sexual Questionnaire (PISQ-12) or Pelvic Organ Prolapse/Urinary Incontinence Sexual Questionnaire, IUGA-Revised (PISQ-IR) | Post-surgery through study completion, approximately 7yrs

CONTACTS AND LOCATIONS:
Overall Officials: Martin Weisberg, MD, Study Director — Ethicon, Inc.
Locations (3):
- United States (2):
  - Institute for Female Pelvic Medicine, North Wales, Pennsylvania
  - UMPC, Pittsburgh, Pennsylvania
- Universitatsklinikum Tubingen, Tübingen, Germany

IPD SHARING:
Plan to Share IPD: Yes
Johnson & Johnson Medical Device Companies have an agreement with the Yale Open Data Access (YODA) Project to serve as the independent review panel for evaluation of requests for clinical study reports and participant level data from investigators and physicians for scientific research that will advance medical knowledge and public health. Requests for access to the study data can be submitted through the YODA Project site at http://yoda.yale.edu.
URL: http://yoda.yale.edu